CLINICAL TRIAL: NCT05537883
Title: Single Blinded Randomized Trial of Transversus Abdominis Plane Block Using Liposomal Bupivacaine in Metabolic and Bariatric Surgery Patients
Brief Title: Transversus Abdominis Plane (TAP) Block Using Liposomal Bupivacaine in Metabolic and Bariatric Surgery Patients
Acronym: TAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00083696
Record Dates: First submitted 2022-09-12; First posted 2022-09-13 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2024-06

CONDITIONS: Morbid Obesity; Bariatric Surgery Candidate
Keywords: Transversus Abdominis Plane (TAP) block; Bupivacaine; Liposomal bupivacaine
MeSH Terms: conditions — Obesity, Morbid; Bites and Stings | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: This study is a 2-arm parallel single blinded randomized equivalency, single-center, clinical trial.
Who Masked: Participant
Masking Description: Patients will be blinded to type of Transversus Abdominis Plane (TAP) block used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine only (Active Comparator): Active control group patients receive Transversus Abdominis Plane (TAP) block with a Bupivacaine only mixture, containing 50 mL 0.5% Bupivacaine, and 100 mL normal saline solution.
  Interventions: Drug: Bupivacaine Injection
- Liposomal Bupivacaine (Experimental): Study group patients will receive Transversus Abdominis Plane (TAP) block with a Liposomal Bupivacaine mixture, containing 20 mL Liposomal Bupivacaine, 30 mL 0.5% Bupivacaine, and 100 mL normal saline solution.
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Patients receiving the intervention will undergo Transversus Abdominis Plane (TAP) block with liposomal bupivacaine
  Other Names: Exparel
  Arms: Liposomal Bupivacaine
Drug: Bupivacaine Injection — Patients receiving the intervention will undergo Transversus Abdominis Plane (TAP) block with plain bupivacaine
  Other Names: Plain bupivacaine
  Arms: Bupivacaine only

SUMMARY:
To investigate if laparoscopic Transversus Abdominis Plane (TAP) block using plain bupivacaine is equivalent to using liposomal bupivacaine in patients undergoing metabolic and bariatric surgery. The study will see if the plain bupivacaine group will be equivalent in terms of length of stay, Morphine Milligram Equivalents, Pain scores and patient satisfaction, but cost less.

DETAILED DESCRIPTION:
Compared to only Bupivacaine administered via TAP block, the study will investigate the analgesia effects to patients undergoing metabolic and bariatric surgery receiving TAP block with a Liposomal Bupivacaine mixture. To determine if patients undergoing metabolic and bariatric surgery receiving TAP block with a Liposomal Bupivacaine results in pain scores, as measured by visual analogic scale (VAS), that are equivalent compared to patients receiving TAP block with Bupivacaine only. Compared to TAP block with Bupivacaine only, the study will compare opioid consumption, and other effect differences to patients undergoing metabolic and bariatric surgery receiving TAP block with Liposomal Bupivacaine. The study will explore other effects, including pain score at 48 hours, and 72 hours after surgery, total opioid consumption required post op during their one-week post op visit as measured in morphine equivalences.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* Participants who can give written informed consent and willing to comply with all study-related procedures.
* Patients undergoing primary sleeve gastrectomy or roux-en-y gastric bypass

Exclusion Criteria:

* Patients undergoing duodenal switch procedures
* Patients undergoing concomitant hiatal hernia repair or ventral hernia repair or cholecystectomy at time of primary metabolic surgery
* Patients with chronic opioid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahman Nimeri, MD, Principal Investigator — Wake Forest University Health Sciences, Atrium Health
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McDonnell JG, O'Donnell BD, Farrell T, Gough N, Tuite D, Power C, Laffey JG. Transversus abdominis plane block: a cadaveric and radiological evaluation. Reg Anesth Pain Med. 2007 Sep-Oct;32(5):399-404. doi: 10.1016/j.rapm.2007.03.011. PMID 17961838
- [Background] Mukhtar K, Singh S. Transversus abdominis plane block for laparoscopic surgery. Br J Anaesth. 2009 Jan;102(1):143-4. doi: 10.1093/bja/aen338. No abstract available. PMID 19059927
- [Background] Hamid HKS, Ahmed AY, Saber AA, Emile SH, Ibrahim M, Ruiz-Tovar J. Transversus abdominis plane block using a short-acting local anesthetic reduces pain and opioid consumption after laparoscopic bariatric surgery: a meta-analysis. Surg Obes Relat Dis. 2020 Sep;16(9):1349-1357. doi: 10.1016/j.soard.2020.04.023. Epub 2020 Apr 24. PMID 32709581
- [Background] Jin Z, Ding O, Islam A, Li R, Lin J. Comparison of Liposomal Bupivacaine and Conventional Local Anesthetic Agents in Regional Anesthesia: A Systematic Review. Anesth Analg. 2021 Jun 1;132(6):1626-1634. doi: 10.1213/ANE.0000000000005406. PMID 33687173
- See also: Patient survey app distribution website — https://seamless.md/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 of the subjects were not randomized or assigned
Period: Overall Study
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine
Started | 35 | 34
Completed | 0 | 0
Not Completed | 35 | 34
Not completed — revisional surgery | 4 | 2
Not completed — surgeries were cancelled | 0 | 2
Not completed — not being compliant with the Seamless MD app | 31 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Customized [Mean (Full Range); unit: Number of years] | 44 [22 to 66] | 43 [23 to 62] | 43.5 [22 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 14 | 29
  White | 19 | 18 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean 24 Hour Visual Analogue Scale (VAS) Pain Score
Description: Pain score at 24 hours post-operative, using visual analogue scale (VAS), ranging from 1 to 10. One indicates no pain, and 10 indicates the worst pain one could imagine.
Time Frame: Hour 24
Population: The numbers analyzed meaning those who received the bupivacaine or not were 35 and 34 However, the Post-Anesthesia Care Unit team nurses did not obtain pain scores on everyone so what is listed is the data of what we had, which is less. This is why it doesn't add up.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 27
score on a scale | 1 [0 to 5] | 3 [0 to 9]

2. Secondary Outcome: Mean Visual Analogue Scale (VAS) Pain Scores
Description: Pain score at 12 hours, 48 hours, and 72 hours post-operative, using visual analogue scale (VAS), ranging from 1 to 10. One indicates no pain, and 10 indicates the worst pain one could imagine
Time Frame: Hours,12, 48, and 72
Population: Difference in Number of Subjects at different Hours due to subjects being non-compliant: not entering information into Seamless MD app; data not being collected The numbers analyzed meaning those who received the bupivacaine or not were 35 and 34 However, the Post-Anesthesia Care Unit team nurses did not obtain pain scores on 6 Subjects in Bupivacaine Group and 7 Subjects in the Liposomal Bupivacaine Group
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine
Number analyzed (Participants) | 29 | 27
score on a scale
  Hour 12: number analyzed (Participants) | 15 | 14
  Hour 12 | 4.4 [0 to 10] | 5.64 [0 to 9]
  Hour 48: number analyzed (Participants) | 10 | 8
  Hour 48 | 5.7 [0 to 9] | 5.6 [2 to 8]
  Hour 72: number analyzed (Participants) | 4 | 5
  Hour 72 | 2.5 [0 to 5] | 7.0 [4 to 8]

3. Secondary Outcome: Mean Average Morphine Equivalences
Description: Morphine milligram equivalences consumed during hospital stay
Time Frame: Day 3
Measure: Mean (Full Range); unit: Morphine Milligram Equivalents
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine
Number analyzed (Participants) | 35 | 34
Morphine Milligram Equivalents
  Intraoperative Administration Bupivacaine: up to 24 hours Liposomal Bupivacaine: up to 25 hours | 11.67 [2 to 24] | 13.1 [10 to 25]
  Post Anesthesia Care Unit (PACU) Bupivacaine: up to 9 hours Liposomal Bupivacaine: up to 6 hours | 4.67 [2 to 9] | 3.43 [2 to 6]
  Floor Admin/Subject Room Bupivacaine: up to 6 hours Liposomal Bupivacaine: up to 22.5 hour | 3.8 [0.8 to 6] | 5.61 [1.6 to 22.5]

4. Secondary Outcome: Morphine Equivalences - Week 1
Description: Morphine milligram equivalences prescribed and consumed as measured at one week follow up clinic visit
Time Frame: Week 1
Population: There were no data points as no patient completed or were non-compliant in completing their Seamless MD Mean Morphine Milligram Equivalents (MME) use and lack of compliance of clinic obtaining this data and submitting into redcap.
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Post-operative Nausea and Vomiting (PONV)
Description: Post-operative nausea and vomiting (PONV) measured by a numerical score (1: no nausea or vomiting, 2: some nausea no vomiting, 3: nausea and vomiting)
Time Frame: Week 1
Population: There were no data points as no patient completed or were non-compliant in completing their Seamless MD MME use and lack of compliance of clinic obtaining this data and submitting into redcap.
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Length of Hospital Stay
Description: Hospital length of stay in hours
Time Frame: Day 3
Measure: Mean (Full Range); unit: hours
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine
Number analyzed (Participants) | 35 | 34
hours | 24.5 [17.5 to 42] | 29.7 [20 to 68]

7. Secondary Outcome: Patient Satisfaction Scores
Description: Patient Satisfaction score based on daily postop online surveys - These parameters will be scored via SeamlessMD on a phone application, as well as paper and pen on a standardized reporting form for patients less comfortable using technology - scored on a scale of 0-10, with 0 being "worst surgeon possible and 10 being "best surgeon possible."
Time Frame: Day 30
Population: as for outcome 5
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Week 1
Description: subjects being non-compliant
Arm/Group | Bupivacaine Only | Liposomal Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 0/35 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/83/NCT05537883/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/83/NCT05537883/ICF_001.pdf